CLINICAL TRIAL: NCT04179877
Title: A Naturalistic Controlled Trial of Individual Placement and Control in Bodø
Acronym: IPSBODO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Nordlandssykehuset HF (Other); University of Tromso (Other); London School of Economics and Political Science (Other); University of Melbourne (Other); St George's Healthcare NHS Trust (Other); The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IPSBODO
Record Dates: First submitted 2018-11-30; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Severe Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Naturalistic controlled trial with one municipality (Bodø) as treatment group and 10 similar municipalities without IPS services as controls.
Masking Description: The control municipalities are unaware of this project, and are thus masked to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual placement and support (Experimental): Group of patients receiving IPS to increase workforce participation.
  Interventions: Behavioral: IPS
- Control (No Intervention): Group of patients receiving treatment as usual.

INTERVENTIONS:
Behavioral: IPS — Occupational rehabilitation and support Integrated with clinical treatment
  Arms: Individual placement and support

SUMMARY:
The investigators aim to test the effectiveness of Individual Placement and Support (IPS) on

1. employment,
2. welfare dependency, and
3. public-sector health care utilization.

This is a naturalistic controlled trial, where one municipality (Bodø in Norway) with about 50000 inhabitants get access to IPS services in public sector mental health services during the period 2013-2016. The target group for the intervention is patients with severe mental illness (SMI) in the age group 18-40 at time of treatment. Patients already receiving lifelong disability benefits will be excluded.

The control group will be an average of 10 municipalities in Norway without IPS services.

Data for outcomes will be based on public registries available for research.

DETAILED DESCRIPTION:
The investigators aim test the hypotheses that Individual Placement and Support (IPS) is effective in

1. increasing employment,
2. reducing welfare dependency, and
3. reducing public-sector health care utilization.

This is a naturalistic controlled trial, where one municipality (Bodø in Norway) with about 50000 inhabitants get access to IPS services in public sector mental health services during the period 2013-2016. The follow-up period will last until 2022. The target group for the intervention is patients with severe mental illness (SMI) in the age group 18-40 at time of treatment, with an ambition of 200 received IPS services. The investigators aim to study the effectiveness on the societal (not individual) level, assuming spill-over effects within Bodø municipality as a result of system changes in the treatment municipality (Bodø). Patients already receiving lifelong disability benefits will be excluded. The control group will be 10 similar municipalities in Norway without IPS services and will be chosen on the basis of similarities in economy, demography and geography and collected from publicly available information. Approximately 77000 subjects will be enrolled in this study; 7000 subjects from Bodø municipality and 70000 from the other 10 municipalities (the control group).

Data for outcomes will be based on public registries available for research. Outcome operationalizations are:

1. Employment will be based on registry data from tax records with information both on employment (yes/no and period) and taxable income (NOK).
2. Welfare dependency will be based on registry data including rehabilitation benefits, disability benefits, sickness absence, unemployment benefits, and social benefits. These will be analysed separate and combined, and the main hypothesis will be based on the latter.
3. Health care utilization will be based on data from the Norwegian Patient Register. Data for in-patient and out-patients treatments for mental illness and other (separate analyses) will be used. These will be analysed separate and combined, and the main hypothesis will be based on the first.

The data will be analyzed in two rounds; first in 2019, and a follow-up analysis in 2022. A difference-in-difference approach will be used to measure the effects.

ELIGIBILITY:
Inclusion Criteria:

* Severe mental illness
* Work assessment allowance

Exclusion Criteria:

* Disability benefit

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Long-term welfare dependency | 15 years after implementation of IPS-services in Bodø (intervention municipality)
  Rates of welfare dependency (rehabilitation benefits, disability benefits, sickness absence, unemployment benefits, and social benefits) in Bodø (intervention municipality) will be compared to rates of welfare dependency in 10 resembling municipalities (Kongsberg, Lier, Røyken, Horten, Tønsberg, Larvik, Færder, Porsgrunn, Grimstad og Steinkjer) without IPS-services (control municipalities) using Norwegian registry data.

SECONDARY OUTCOMES:
Employment rate | 3 years after implementation of IPS-services in Bodø, Norway
  Rates of employment in Bodø (intervention municipality) will be compared to employment rates in 10 resembling municipalities (Kongsberg, Lier, Røyken, Horten, Tønsberg, Larvik, Færder, Porsgrunn, Grimstad og Steinkjer) without IPS-services (control municipalities). The measurement tool will be Norwegian registry data from tax records with information both on employment (yes/no and time period) and taxable income (NOK).
Employment rate | 7 years after implementation of IPS-services in Bodø, Norway (intervention municipality)
  Rates of employment in Bodø (intervention municipality) will be compared to employment rates in 10 resembling municipalities (Kongsberg, Lier, Røyken, Horten, Tønsberg, Larvik, Færder, Porsgrunn, Grimstad og Steinkjer) without IPS-services (control municipalities). The measurement tool will be Norwegian registry data from tax records with information both on employment (yes/no and time period) and taxable income (NOK).
Welfare dependency rate | 3 years after implementation of IPS-services in Bodø (intervention municipality)
  Welfare dependency rates (rehabilitation benefits, disability benefits, sickness absence, unemployment benefits, and social benefits) in Bodø (intervention group/municipality) will be compared to 10 similar municipalities without IPS-services (control groups/municipalities).
Welfare dependency rate | 7 years after implementation of IPS-services in Bodø (intervention municipality)
  Rates of welfare dependency (rehabilitation benefits, disability benefits, sickness absence, unemployment benefits, and social benefits) in Bodø (intervention municipality) will be compared to rates of welfare dependency in 10 resembling municipalities (Kongsberg, Lier, Røyken, Horten, Tønsberg, Larvik, Færder, Porsgrunn, Grimstad og Steinkjer) without IPS-services (control municipalities) using Norwegian registry data.
Rates of treatments for mental illness | 3 years after implementation of IPS-services in Bodø (intervention municipality)
  Rates of health care utilization in Bodø (intervention municipality) will be compared to health care utilization rates in 10 resembling municipalities (Kongsberg, Lier, Røyken, Horten, Tønsberg, Larvik, Færder, Porsgrunn, Grimstad og Steinkjer) without IPS-services (control municipalities). Health care utilization will be based on data from the Norwegian Patient Register. We will use data for in-patient and out-patients treatments for mental illness and other (separate analyses), collected from the Norwegian Patient Register as a measurement tool. These will be analysed separate and combined, and the main hypothesis will be based on the first.
Rates of treatments for mental illness | 7 years after implementation of IPS-services in Bodø (intervention municipality)
  Rates of health care utilization in Bodø (intervention municipality) will be compared to health care utilization rates in 10 resembling municipalities (Kongsberg, Lier, Røyken, Horten, Tønsberg, Larvik, Færder, Porsgrunn, Grimstad og Steinkjer) without IPS-services (control municipalities). Health care utilization will be based on data from the Norwegian Patient Register. We will use data for in-patient and out-patients treatments for mental illness and other (separate analyses), collected from the Norwegian Patient Register as a measurement tool. These will be analysed separate and combined, and the main hypothesis will be based on the first.

CONTACTS AND LOCATIONS:
Overall Officials: Arnstein Mykletun, Prof PsyD, Principal Investigator — Norwegian IPH
Locations (1):
- Nordland Hospital Trust, Bodø, Nordland, Norway

IPD SHARING:
Plan to Share IPD: No